CLINICAL TRIAL: NCT03187964
Title: Feasibility, Accuracy, and Effect of Polyvalent Point-of-care Xpert MTB/RIF Ultra and Xpert HIV-1 Viral Load Testing in HIV-positive Patients Initiating ART: a Randomised Controlled Trial
Brief Title: Xpert Ultra and Xpert HIV-VL in People Living With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Stellenbosch (Other)
Responsible Party: Principal Investigator, Grant Theron, Associate Professor, University of Stellenbosch
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: N14/10/136
Record Dates: First submitted 2017-06-12; First posted 2017-06-15 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: HIV/AIDS; TB - Tuberculosis; Antiretroviral Therapy, Highly Active
Keywords: People Living with HIV (PLHIV); Xpert HIV-1 Viral Load (Xpert VL); Xpert Ultra; Antiretroviral treatment (ART)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Latent Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PLHIV Centralised Xpert Ultra (No Intervention): Patient sputum specimen collected at Kraaifontein Community Health Centre (KCHC) and sent for centralised Xpert Ultra TB testing at the National Health Laboratory Services (NHLS) facility in Greenpoint, Cape Town, South Africa. Centralised testing uses the established NHLS transportation, testing and report-back to clinic infrastructure according to the national algorithm.
- PLHIV Point of Care Xpert Ultra (Active Comparator): Patient sputum specimen collected at KCHC and Xpert Ultra TB testing done on site at point of care (POC).
  Interventions: Diagnostic Test: PLHIV Point of Care Xpert Ultra
- PLHIV Centralised Xpert VL (No Intervention): Patient blood specimen collected at Kraaifontein Community Health Centre (KCHC) and sent for centralised viral load testing at the NHLS facility in Tygerberg Hospital, Cape Town, South Africa. Centralised testing uses the established NHLS transportation, testing and report-back to clinic infrastructure according to the national algorithm.
- PLHIV Point of Care Xpert VL (Active Comparator): Patient blood specimen collected at KCHC and Xpert HIV-1 viral load testing done on site at point of care (POC).
  Interventions: Diagnostic Test: PLHIV Point of Care Xpert VL

INTERVENTIONS:
Diagnostic Test: PLHIV Point of Care Xpert Ultra — Sputum-based TB diagnostic test that takes 80 min to run. Test performed on the same day as the patient visit.
  Other Names: GeneXpert
  Arms: PLHIV Point of Care Xpert Ultra
Diagnostic Test: PLHIV Point of Care Xpert VL — Blood-based HIV-1 VL diagnostic and monitoring test that takes 60 min to run. Test performed on the same day as the patient visit.
  Other Names: GeneXpert
  Arms: PLHIV Point of Care Xpert VL

SUMMARY:
TB is increasingly diagnosed using the GeneXpert platform, which can be used for a variety of tests (not just TB). HIV viral load monitoring is required at least annually in patients on ART to detect failure of virologic suppression, however, most HIV VL testing is done centrally. A patient with virologic failure is more likely to get TB.

The investigators wish to see if Xpert done at the clinic results in faster patient TB diagnosis and treatment initiation compared to sending specimens away for central testing. In a different patient group (PLHIV returning for HIV treatment monitoring), the investigators wish to see if POC Xpert HIV-1 viral load (Xpert VL) testing results in faster patient viral load quantification compared to centralised testing. Both POC tests will use the same testing hardware. This polyvalent utility of the GeneXpert system is hitherto uninvestigated in this local setting.

Newly diagnosed pre-ART HIV positive patients will be approached and asked to be a part of this study. Patients will be randomly assigned to Ultra done at the clinic or the normal off-site laboratory TB testing. The time taken for patients to get diagnosed and time-to-treatment will be recorded. We will also do exploratory diagnostic accuracy evaluations including but not limited to, Ultra when done on mouth samples, the new SILVAMP FujiLAM on urine, and host RNA blood signatures for active TB. Additionally, a different group of HIV positive patients (on ART) returning to the clinic for annual follow-up visits will also be asked to join the study. These patients will be randomly selected for either Xpert VL testing done at the clinic or the normal off-site testing. The time taken for patients to receive viral load results will be recorded. Should the patient's viral loads be found to be higher than anticipated and considered by the clinical to indicate a lack of viral suppression, the time taken for patients to have ART regimen adjusted, receive adherence counselling or received HIV drug susceptibility testing will be recorded.

This project will confirm if Ultra TB testing performs well in PLHIV irrespective of symptoms and may produce evidence that supports universal TB testing in this important and vulnerable patient group, including using novel diagnostics on non-traditional specimen types. The investigators will also assess whether POC placement of Ultra and Xpert VL has benefits (e.g., more patients diagnosed for TB or VL monitored during the same day visit).

DETAILED DESCRIPTION:
Sensitive and rapid point-of-care diagnostics should improve TB treatment outcomes, however, tests meeting these criteria have, until recently, been unavailable, especially in PLHIV. PLHIV often have early stage TB disease at the time of ART initiation and paucibacillary sputum. The current frontline test for TB is the Xpert MTB/RIF, which uses the GeneXpert platform, and is deployed primarily at centralised reference laboratories (Clouse et al., 2012; Hanrahan et al., 2015). This approach has two major limitations: 1) the instruments' far-patient placement likely undermines its potential clinical impact; 2) Xpert MTB/RIF has suboptimal sensitivity in PLHIV 3) the GeneXpert platform is primarily used only for TB testing and no other assays such as Xpert HIV-1 Viral Load (VL).

Xpert MTB/RIF has been succeeded by Xpert MTB/RIF Ultra (Xpert Ultra), which promises to increase the speed and sensitivity of TB diagnosis. Although Xpert Ultra will doubtlessly improve the detection of symptomatic patients, its greatest incremental benefit will likely arise in patients with low bacillary load (e.g., unselected HIV-positive patients initiating ART). Thus, Xpert Ultra has the potential to alter how TB is diagnosed in PLHIV by detecting TB before the disease has a chance to progress and before substantial transmission has occurred. The investigators will, in addition to Xpert Ultra on sputum, also perform TB testing using the urinary lateral flow (LF) LAM test, which may detect mycobacteria in asymptomatic PLHIV patients (Lawn et al., 2011). Moreover, investigators will also perform Xpert Ultra and Fujifilm SILVAMP (FujiLAM) on urine in ART initiators. Oral sampling will be done which includes the use of Ultra on tongue swabs and oral washes, inhouse PCR testing MGIT960 liquid culture from PLHIV (ART initiators) as part of preliminary investigation will also be explored, as well the use of blood RNA signatures for TB diagnosis.

These novel test investigations are exploratory, and the results will not yet be used for patient management. This study will address the following research questions: (1) What is the sensitivity and specificity for each approach, overall, and after stratification by viral load/CD4, and (2) What is the proportion of patients that could not expectorate sputum were detected by non-sputum based tests?

The polyvalent utility of the GeneXpert hardware platform is, however, hitherto largely unexplored despite the widespread deployment of machines. HIV VL testing is currently done in South Africa according to the National HIV Treatment guidelines, which advise measuring HIV VL every six months for the first year of treatment and annually thereafter. HIV VL testing involves collection of a blood sample, transporting it to a centralised laboratory for VL quantification, reporting the result back to the clinic, and calling the patient back. If HIV VL is found to be over 1000 genomes per ml, the patient may not be adherent to the prescribed ART or may have drug-resistant HIV and, now that a failure of virologic suppression has been confirmed, the patient may be asked to give a second blood sample for drug susceptibility testing and may have a counselling visit scheduled, in order to improve the patient's adherence. There is, however, a large amount of discretion at local clinics as to what constitutes virologic failure and patients with increased VL may still receive these interventions, even if below the 1000 genomes per ml threshold. The investigators also intend to perform Xpert HIV-1 VL testing and, compared to patients who receive the standard-of-care of centralised VL testing, evaluate the proportion of patients without virologic suppression who are referred to a follow-up intervention (DST and/or adherence counselling).

The investigators propose a study which implements Xpert Ultra (in unselected PLHIV) and Xpert HIV-1 VL (in PLHIV on ART) in Cape Town, South Africa. Furthermore, the GeneXpert platform's polyvalent feasibility, time-to-result and -treatment (Xpert Ultra and LF LAM), and effect on interventions to improve VL (Xpert HIV-1 VL) will be examined.

ELIGIBILITY:
HIV-positive viral load monitoring patients

Inclusion Criteria:

* Informed consent obtained from patient
* Patient is more than 18 years old
* Patient is HIV positive
* Patient is receiving follow-up ART
* Patient is willing to provide blood specimens for study

Exclusion Criteria:

* Informed consent not obtained from patient
* Patient is less than 18 years old
* Patient is HIV negative or has unknown HIV status
* Patient is coming into clinic for first time ART
* Patient is not willing to provide blood specimens for study

TB patients

Inclusion Criteria:

* Informed consent obtained from patient
* Patient is more than 18 years old
* Patient is HIV positive
* Patient is coming into clinic for first ART visit
* Patient is willing to provide sputum and urine (blood is desirable, but not mandatory) specimens for study

Exclusion Criteria:

* Informed consent not obtained from patient
* Patient is less than 18 years old
* Patient is HIV negative or has unknown HIV status
* Patient is not coming into clinic for first time ART
* Patient has been on TB treatment within the last 60 days
* Patient is not willing to provide sputum and urine specimens for study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1053 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2022-01-16 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Treatment time | Up to 8 weeks
  Time-specific proportion of patients starting TB treatment (all patients and confirmed cases) in centralised diagnosis and treatment arm compared to POC arm (Xpert Ultra).

SECONDARY OUTCOMES:
TB diagnosis time | Up to 8 weeks
  Time-specific proportion of patients diagnosed in centralised diagnosis and treatment arm compared to POC arm (Xpert Ultra for TB and XpertVL for VL)
Urine LF-LAM, urine FujiLAM and urine Xpert Ultra in people investigated for TB | Up to one week
  Diagnostic accuracy and concordance compared to a sputum culture reference standard
Tongue swab and oral wash Xpert Ultra, tongue swab in-house PCR, and tongue swab culture in people investigated for TB | Up to one week
  Diagnostic accuracy and concordance compared to a sputum culture reference standard and vs. the tongue swab culture
Candidate host RNA blood signatures for active TB specified in Turner LRM et al., 2020 in people investigated for TB | Up to one week
  Diagnostic accuracy and concordance compared to a sputum culture reference standardUU
HIV DST or adherence counselling | Up to one week
  Time-specific proportion of patients without virologic suppression identified to require adherence counselling and/or HIV drug susceptibility testing
Time to referral for HIV regimen adjustment or adherence counselling in patients without virologic suppression | Up to 8 weeks
  Time-specific proportion of patients without virologic suppression referred for adherence counselling and/or switching to a second-line ART regimen
Initial lost to follow-up | Up to 12 weeks
  Time-specific proportion of patients with a known TB diagnosis or increase in HIV VL that do not successfully start treatment (TB) or HIV adherence counselling, DST or regimen change (VL)

CONTACTS AND LOCATIONS:
Overall Officials: Grant Theron, PhD, Principal Investigator — University of Stellenbosch
Locations (1):
- Kraaifontein Community Health Centre, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Collaborators will have access to de-identified IPD data. Other researchers wishing to access the data will be required to sign a data sharing agreement as per institutional policies.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be available once the findings are published.
Access Criteria: Data access will be granted to interested collaborators and parties through sharing of data files or login information for the study's secure RedCap electronic database during the course of patient recruitment.

REFERENCES:
- [Background] Hanrahan CF, Clouse K, Bassett J, Mutunga L, Selibas K, Stevens W, Scott L, Sanne I, Van Rie A. The patient impact of point-of-care vs. laboratory placement of Xpert((R)) MTB/RIF. Int J Tuberc Lung Dis. 2015 Jul;19(7):811-6. doi: 10.5588/ijtld.15.0013. PMID 26056107
- [Background] Lawn SD, Brooks SV, Kranzer K, Nicol MP, Whitelaw A, Vogt M, Bekker LG, Wood R. Screening for HIV-associated tuberculosis and rifampicin resistance before antiretroviral therapy using the Xpert MTB/RIF assay: a prospective study. PLoS Med. 2011 Jul;8(7):e1001067. doi: 10.1371/journal.pmed.1001067. Epub 2011 Jul 26. PMID 21818180
- [Background] Clouse K, Page-Shipp L, Dansey H, Moatlhodi B, Scott L, Bassett J, Stevens W, Sanne I, Van Rie A. Implementation of Xpert MTB/RIF for routine point-of-care diagnosis of tuberculosis at the primary care level. S Afr Med J. 2012 Sep 7;102(10):805-7. doi: 10.7196/samj.5851. PMID 23034211
- [Background] Luabeya AK, Wood RC, Shenje J, Filander E, Ontong C, Mabwe S, Africa H, Nguyen FK, Olson A, Weigel KM, Jones-Engel L, Hatherill M, Cangelosi GA. Noninvasive Detection of Tuberculosis by Oral Swab Analysis. J Clin Microbiol. 2019 Feb 27;57(3):e01847-18. doi: 10.1128/JCM.01847-18. Print 2019 Mar. PMID 30541931
- [Background] Broger T, Sossen B, du Toit E, Kerkhoff AD, Schutz C, Ivanova Reipold E, Ward A, Barr DA, Mace A, Trollip A, Burton R, Ongarello S, Pinter A, Lowary TL, Boehme C, Nicol MP, Meintjes G, Denkinger CM. Novel lipoarabinomannan point-of-care tuberculosis test for people with HIV: a diagnostic accuracy study. Lancet Infect Dis. 2019 Aug;19(8):852-861. doi: 10.1016/S1473-3099(19)30001-5. Epub 2019 May 30. PMID 31155318
- [Background] Turner CT, Gupta RK, Tsaliki E, Roe JK, Mondal P, Nyawo GR, Palmer Z, Miller RF, Reeve BW, Theron G, Noursadeghi M. Blood transcriptional biomarkers for active pulmonary tuberculosis in a high-burden setting: a prospective, observational, diagnostic accuracy study. Lancet Respir Med. 2020 Apr;8(4):407-419. doi: 10.1016/S2213-2600(19)30469-2. Epub 2020 Mar 13. PMID 32178775
- [Derived] Zifodya JS, Kreniske JS, Schiller I, Kohli M, Dendukuri N, Schumacher SG, Ochodo EA, Haraka F, Zwerling AA, Pai M, Steingart KR, Horne DJ. Xpert Ultra versus Xpert MTB/RIF for pulmonary tuberculosis and rifampicin resistance in adults with presumptive pulmonary tuberculosis. Cochrane Database Syst Rev. 2021 Feb 22;2(2):CD009593. doi: 10.1002/14651858.CD009593.pub5. PMID 33616229